CLINICAL TRIAL: NCT00465374
Title: A Validation/Interventional Study on Stress Index in Predicting Mechanical Stress in ARDS Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRN60ANRA04
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: ARDS; Pressure/time curve; Stress Index
MeSH Terms: conditions — Respiratory Distress Syndrome

INTERVENTIONS:
Procedure: Change ventilatory parameters with stress index monitoring

SUMMARY:
30% of ARDS patients ventilated according to NIH protocol presents CT scan evidence of hyperinflation. Functional analysis of pressure-time curve (Stress Index=SI) has been shown to identify this condition in experimental settings. We tested the hypothesis that the SI is an accurate predictor of mechanical stress due to overdistention in ARDS patients.

DETAILED DESCRIPTION:
The study presents two parts : a preliminary validation study and a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of ARDS based on American-European Consensus Conference criteria

Exclusion Criteria:

* >3 days since ARDS criteria were met and mechanical ventilation was started
* History of ventricular fibrillation or tachyarrhythmia, unstable angina or myocardial infarction within preceding month
* Pre-existing chronic obstructive pulmonary disease
* Major chest wall abnormalities
* Chest tube with persistent air leak
* Abdominal distension
* Body mass index >30
* Pregnancy
* Known intracranial abnormality
* Enrollment in another interventional study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10

PRIMARY OUTCOMES:
reduction of pulmonary inflammatory mediators

CONTACTS AND LOCATIONS:
Overall Officials: V. M. Ranieri, MD, Study Director — University of Turin, Italy; P. Terragni, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- University of Turin, Department of Anesthesia and Intensive Care Medicine, Turin, Italy

REFERENCES:
- [Background] Ranieri VM, Zhang H, Mascia L, Aubin M, Lin CY, Mullen JB, Grasso S, Binnie M, Volgyesi GA, Eng P, Slutsky AS. Pressure-time curve predicts minimally injurious ventilatory strategy in an isolated rat lung model. Anesthesiology. 2000 Nov;93(5):1320-8. doi: 10.1097/00000542-200011000-00027. PMID 11046222
- [Background] Grasso S, Terragni P, Mascia L, Fanelli V, Quintel M, Herrmann P, Hedenstierna G, Slutsky AS, Ranieri VM. Airway pressure-time curve profile (stress index) detects tidal recruitment/hyperinflation in experimental acute lung injury. Crit Care Med. 2004 Apr;32(4):1018-27. doi: 10.1097/01.ccm.0000120059.94009.ad. PMID 15071395